CLINICAL TRIAL: NCT07252232
Title: RASolute 304: A Phase 3 Multicenter, Open-label, Randomized, 2-Arm Study of Adjuvant Daraxonrasib Versus Standard of Care Observation Following Completion of Neoadjuvant and/or Adjuvant Chemotherapy in Patients With Resected Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: Study of Daraxonrasib (RMC-6236) in Patients With Resected Pancreatic Ductal Adenocarcinoma (PDAC)
Acronym: RASolute 304
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-6236-304
Record Dates: First submitted 2025-11-13; First posted 2025-11-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer; PDAC; PDAC - Pancreatic Ductal Adenocarcinoma; Resectable Pancreatic Ductal Adenocarcinoma (PDAC); Resected Pancreatic Adenocarcinoma
Keywords: Pancreatic Cancer; PDAC; Pancreatic Ductal Adenocarcinoma; RAS; KRAS; NRAS; HRAS; RAS Wild-Type; RASolute; Resectable Pancreatic Ductal Adenocarcinoma; Resectable PDAC; Resected Pancreatic Adenocarcinoma; RAS Mutation
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- daraxonrasib (Experimental): study drug
  Interventions: Drug: daraxonrasib
- SOC Observation (No Intervention): Patients randomized to the comparator control arm will receive SOC observation.

INTERVENTIONS:
Drug: daraxonrasib — oral tablets
  Arms: daraxonrasib

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a novel RAS(ON) inhibitor compared to standard of care (SOC) observation only.

DETAILED DESCRIPTION:
This is a global, randomized, open-label, Phase 3 study designed to evaluate whether treatment with daraxonrasib will improve disease-free survival (DFS) compared to SOC observation in patients with resected PDAC who have completed neoadjuvant and/or adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and has provided informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Histologically confirmed PDAC with successful (R0/R1) curative intent surgical resection and no evidence of recurrent or metastatic disease.
* Must have received perioperative (neoadjuvant, adjuvant, or a combination of both) multi-agent chemotherapy.
* Must have completed most recent treatment within the past 12 weeks.
* Adequate organ function (bone marrow, liver, kidney, coagulation).
* Documented RAS mutation status.
* Able to take oral medications.

Exclusion Criteria:

* Prior therapy with direct RAS-targeted therapy (eg. degraders and/or inhibitors).
* Any conditions that may affect the ability to take or absorb study drug.
* Major surgery within 28 days prior to randomization.
* Patient is unable or unwilling to comply with protocol-required study visits or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2029-05-10 (Estimated); Study Completion 2030-07-10 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) per Investigator | Up to approximately 5 years
  DFS defined as the time from randomization until disease recurrence or death from any cause, whichever occurs first. Recurrence is per response evaluation criteria in solid tumors (RECIST) v1.1 as assessed by Investigator.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization until death from any cause.
DFS per blinded independent central review (BICR) | Up to approximately 5 years
  DFS defined as the time from randomization until disease recurrence or death from any cause, whichever occurs first. Recurrence is per RECIST v1.1 as assessed by BICR.
DFS Rate at 1 year and 2 years | Up to approximately 2 years
  DFS rate defined as percentage of patients who are disease free at 1 year and 2 years, respectively.
OS rate at 1 year and 2 years | Up to approximately 2 years
  OS rate defined as percentage of patients who are alive at 1 year and 2 years, respectively.
Safety and tolerability of daraxonrasib | Up to approximately 5 years
  Incidence of adverse events (AEs) and changes from baseline in vital signs, ECOG performance score, and clinical laboratory tests.
Pharmacokinetics (PK) | Up to Cycle 4 Day 1 (Day 85)
  Predose concentration of daraxonrasib

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Hartford Healthcare, Hartford, Connecticut
  - Community Health Network, Indianapolis, Indiana
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Taylor Cancer Research Center, Maumee, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Virginia Cancer Specialists, Fairfax, Virginia
- Pan American Oncology Trials, LLC, San Juan, Puerto Rico, Puerto Rico